CLINICAL TRIAL: NCT07126535
Title: Assessment of Esophageal Distensibility and Mucosal Impedance in Dysplastic Barrett's Esophagus Patients Undergoing Radiofrequency Ablation
Brief Title: Impact of RFA on Esophageal Distensibility and Mucosal Impedance
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 25-004350; NCI-2025-05191 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Dysplastic Barrett's Esophagus; Radiofrequency Ablation; Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Esophageal biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Radiofrequency ablation alone — If there is no evidence of nodularity, these patients will undergo RFA. Clinical biopsies utilizing a large-capacity biopsy forceps (Radial Jaw 4, Boston Scientific, Marlborough, MA) are obtained. RFA may be delivered through several devices under the BarrX RFA System (Medtronic USA, Minnetonka, MN), including a circumferential balloon catheter (Halo 360; figure 1), or over the scope focal catheter (Halo 90 or 60). The Halo 360 treats a circumferential 4 cm segment at a time, whereas the focal catheters treat a 1.3x2 cm (Halo 90) or 1.0x1.5 cm (Halo 60) area.

SUMMARY:
Patients undergoing ablative therapy for management of dysplastic Barrett's Esophagus (BE) will have decreased distensibility over the course of treatment, but improvement in mucosal impedance as BE epithelia is replaced by neosquamous epithelia. This information may lead to further research in predicting therapeutic response and complications. The purpose of this research is to collect information while measuring changes related to the esophagus in patients that receive radiofrequency ablation (RFA) for dysplastic Barrett's Esophagus (BE) or esophageal cancer. Study participation includes measurements of the esophagus with the use of two different devices. This takes place during clinically indicated upper endoscopies during the timeframe the participant is receiving RFA treatments. This process will take up to an additional 10 minutes during the upper endoscopy and be done while the participant is sedated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Confirmed histologic diagnosis of BE with dysplasia or intramucosal carcinoma (IMCa)
* Ability to take high-dose proton pump inhibitor (PPI) therapy (such as omeprazole 40 mg BID)
* Willing to undergo multiple rounds of endoscopic eradication therapy (EET) for management of BE (which is the guideline clinical recommendation for management of this disease)

Exclusion Criteria:

* History of esophageal ablation
* History of esophageal stricture
* History of esophageal or gastric surgery
* Pregnancy
* History of achalasia
* History of delayed gastric emptying confirmed by 4-hour gastric emptying study
* Receipt of glucagon-like peptide-1 agonists
* Adults lacking the capacity to consent for self
* Lack of English fluency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the Mayo Clinic Rochester Barrett's Esophagus practice. Clinic and upper endoscopy lists will be screened on a daily basis to identify patients who meet inclusion criteria. These patients will then be invited to participate in the study and screened by the study team.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Changes in distensibility index (DI) | Every 12 weeks, up to 1 year (4 visits)
  Change in DI will be measured by functional luminal impedance planimetry (FLIP) during RFA procedure.
Changes in diameter | Every 12 weeks, up to 1 year (4 visits)
  Change in esophageal diameter will be measured by functional luminal impedance planimetry (FLIP) during RFA procedure.

SECONDARY OUTCOMES:
Changes in mucosal impedance | Every 12 weeks, up to 1 year (4 visits)
  Damage to the mucosal lining of the esophagus and measurement of esophageal leakiness will be assessed by sensors used during RFA procedure.

OTHER OUTCOMES:
GERD-Q Questionnaire | Every 12 weeks, up to 1 year (4 visits)
  The Gastroesophageal Reflux Disease Questionnaire (GERD-Q) IS a 6-item questionnaire used to help diagnose GERD and assess the impact of symptoms on a patient's daily life. Scores range from 0-18 with higher scores indicating greater GERD symptoms.
Reflux symptom index (RSI) | Every 12 weeks, up to 1 year (4 visits)
  The RSI is used to measure impact of GERD symptoms over the past month. It consists of 9 symptoms which are rated on a scale of 0-5 where 0=no problem and 5=significant problem. Higher scores indicate greater impact of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Chamil C Codipilly, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials